CLINICAL TRIAL: NCT03975907
Title: Open Label, Phase I/II Clinical Trial to Evaluate the Safety and Efficacy of Fully Human Anti-BCMA Chimeric Antibody Receptor Autologous T Cell （CAR T）in Patients With Relapsed and/or Refractory Multiple Myeloma (LUMMICAR STUDY 1)
Brief Title: Clinical Trial to Evaluate CT053 in Patients With Relapsed and/or Refractory Multiple Myeloma (LUMMICAR STUDY 1)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CARsgen Therapeutics Co., Ltd. (Industry)
Collaborators: Beijing Chao Yang Hospital (Other); The First Affiliated Hospital of Soochow University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Tianjin Medical University General Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Beijing Hospital (Other Government); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Xiangya Hospital of Central South University (Other); Peking University People's Hospital (Other); Qilu Hospital of Shandong University (Other); Sun Yat-sen University (Other); First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT053-MM-01
Record Dates: First submitted 2019-05-30; First posted 2019-06-05 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; car-T
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Phase I is an open-label, dose escalation study and 2 cohorts to evaluate the safety and tolerability of treatment with CT053 and to determine maximum tolerable dose (MTD) and the Recommended Phase 2 Dose (RP2D) for CT053.
  Phase 2 is a single-arm, open, multi-center study, to evaluate the efficacy and safety of CAR-BCMA T cells (CT053) in subjects with RR/MM.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-BCMA T Cells (Experimental): Phase I: The subjects are enrolled into 2 dose level cohorts in sequence. Phase II: Single arm
  Interventions: Biological: CAR-BCMA T Cells

INTERVENTIONS:
Biological: CAR-BCMA T Cells — The CAR-BCMA T cells (study drug) used in this study are chimeric antigen receptor specifically expressing T cells targeting BCMA.

SUMMARY:
This is an open-label, single arm study to evaluate the safety and tolerability of treatment with CT053 CAR-BCMA T in patients with relapsed and/or refractory multiple myeloma.

DETAILED DESCRIPTION:
The study is composed of two stages, Phase I stage is for dose escalation and recommendation of phase 2 dose, and Phase II stage is to Detailed Description: verify the efficacy and safety of the dose proposed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients and legally acceptable representative must have voluntarily signed ICF and willing to complete the study procedure, after fully understanding of the study.
2. Age ≥ 18 years and ≤ 75 years, male or female
3. The patients have received at least 3 prior lines for MM, (Induction therapy followed by autologous transplantation[ASCT] and maintenance therapy represents one line of therapy, those who have not been treated with ASCT should have documented rationale); For each line of therapy, the patient should have received at least one standard treatment cycle (2016 IMWG) unless the best response to the treatment line is documented as progressive diseases (PD)
4. The patients should have received treatment with at least one proteasome inhibitor AND one immunomodulatory drug, and have ever been relapsed or deteriorated after treatment with at least one regimen consisting of above-mentioned medications (combination or single use)；
5. Patient should be relapsed within 12 months after the last line of therapy, or disease progressed within 60 days after last line of therapy (IMWG criteria 2016), with documented evidence.
6. The patients should have measurable disease based on at least one of the following parameters：

   * Serum M-protein ≥ 10 g/L;
   * Urine M-protein ≥ 200 mg/24 hrs;
   * For those whose Serum or Urine M- protein dose not meed the measurable criteria but the light chain type, serum free light chain (FLC): involved FLC level ≥ 10 mg/dL (100 mg/L) provided serum FLC ratio is abnormal
7. Estimated life expectancy > 12 weeks
8. ECOG performance score 0-1；
9. Sufficient venous access for leukapheresis collection, and no other contraindications to leukapheresis
10. Patients should maintain adequate organ function
11. Women of childbearing age must undergo a serum pregnancy test with negative results before screening and lymphodepletion preconditioning with fludarabine and cyclophosphamide, and are willing to use effective and reliable method of contraception for at least 1 year after T cell infusion
12. Men who actively have intercourse with child-bearing potential women must be willing to use effective and reliable method of contraception for at least 1 year after T cell infusion

Exclusion Criteria:

1. Pregnant or lactating women；
2. Positive for any following tests: human immunodeficiency virus (HIV) antibody, Treponema Pallidum antibody, hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg), HBV e antigen (HBeAg), HBV e antibody, hepatitis B core antibody, HBV DNA;
3. Patients with any uncontrolled active infection including but not limited to active tuberculosis.
4. Patients with AEs from previous treatment that have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) ≤ 1, excluding hair loss, neuropathy and other events that the treating physician can determine to be tolerable.
5. Patients who have ever had any CAR T cell therapy；
6. Patients who have ever had anti-BCMA therapy；
7. Patients have received allogeneic stem cell transplantation for treating multiple myeloma;
8. Patients have received autologous stem cell transplantation less than 12 weeks before leukapheresis；
9. Patients have received any anti-cancer treatment within 14 days before leukapheresis including but not limited to cytotoxic therapy, proteasome inhibitors, immunomodulatory agents, targeted therapies, epigenetic therapy or experimental drug therapy. If the field of radiation covers ≤ 5% of the bone marrow, the subjects are eligible to participate in the study regardless of the radiotherapy end date；
10. Patients have received ≥ 5 mg prednisone daily or other equivalent dose of steroids within 14 days before leukapheresis or lymphodepletion；
11. Patients have plasma cell leukemia, Waldenström macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes) syndrome or AL amyloidosis；
12. Patients have been administered live attenuated vaccine 4 weeks before leukapheresis or lymphodepletion
13. Patients allergic to component of study treatment.
14. Patients have any of the condition as following within 6 months of ICF sign-off: New York Heart Association (NYHA) stage III or IV congestive heart failure, angina pectoris, myocardial infarction, coronary artery bypass graft, stroke (excluding lacunar stroke), history of clinically significant arrhythmia including but not limited to ventricular arrhythmia, significant QT interval prolongation, uncontrolled blood pressure as defined as systolic > 160 mmHg, diastolic > 100 mmHg, uncontrolled diabetes mellitus, pulmonary thrombolism, other conditions that investigators believe that participating in this clinical trial may endanger the health of the patients
15. Patients are known to have active autoimmune diseases including but not limited to psoriasis, rheumatoid arthritis and other needs of long-term immunosuppressive therapy
16. patients are oxygen dependent as defined by the blood oxygen saturation (finger oxygen detection method) can be maintained > 95% only by oxygen inhalation before leukapheresis
17. Patients with second malignancies in addition to MM are not eligible if the second malignancy has required treatment within the past 5 years or is not in complete remission. There are two exceptions to this criterion: successfully treated cervical carcinoma in situ and non-metastatic basal cell skin carcinoma
18. Patients have central nervous system (CNS) metastases or CNS involvement (including cranial neuropathies or mass lesions and leptomeningeal disease). Patients with history of spinal cord compression from MM are eligible provided spinal cord compression has been treated with surgery or radiation at least 28 days prior to study entry
19. Patients are unable or unwilling to comply with the requirements of clinical trial
20. Patients have received major surgery 2 weeks prior to leukapheresis or 4 weeks prior to lymphodepletion and after the study treatment (excluding cataract and other local anesthesia)
21. Patients are relatives to investigator or his/her staff, or those who may have an interest in the investigator and/or his/her staff.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1, Safety and tolerability: dose limiting toxicity | 28days post administration of CAR-T-cells
  dose limiting toxicity
Phase 2, efficacy of CT053 CAR-BCMA T cells: overall response rate | 3 months post administration of CAR-T-cells
  overall response rate (ORR)=（sCR+CR+VGPR+PR)

SECONDARY OUTCOMES:
Additional efficacy evaluation after 12 weeks of CT053 CAR-BCMA T cells infusion | 3 months post administration of CAR-T-cells
  Minimal residual disease (MRD) negativity
Additional efficacy evaluation after 12 weeks of CT053 CAR-BCMA T cells infusion | 3 months post administration of CAR-T-cells
  TTR TIme to Response
Additional efficacy evaluation after 12 weeks of CT053 CAR-BCMA T cells infusion | 3 months post administration of CAR-T-cells
  Complete Response (CR) /stringent Complete Response (sCR)
Additional efficacy evaluation after 12 weeks of CT053 CAR-BCMA T cells infusion | 3 months post administration of CAR-T-cells
  ≥Very Good Partial Response (VGPR), including VGPR, CR, sCR
Additional efficacy evaluation after 12 weeks of CT053 CAR-BCMA T cells infusion | 3 months post administration of CAR-T-cells
  ORR at Wk12
Additional efficacy evaluation after 12 weeks of CT053 CAR-BCMA T cells infusion | 3 months post administration of CAR-T-cells
  CBR, clinical benefit rate
Safety and tolerability of CAR-BCMA T cell therapy | through 24 months post administration of CAR-T-cells
  AE&SAE
Pharmacokinetics (the cell persistence duration in peripheral blood) | through 24 months post administration of CAR-T-cells
  Copy numbers of CAR-BCMA gene in peripheral blood
Pharmacokinetics (the cell persistence duration in peripheral blood) | through 24 months post administration of CAR-T-cells
  Number of CAR positive cells in peripheral blood
Safety and tolerability of CAR-BCMA T cell therapy | through 24 months post administration of CAR-T-cells
  positivity of ADA (Anti-CAR-T antibody)
Efficacy endpoint of CAR-BCMA T cells after infusion | through 24 months post administration of CAR-T-cells
  Overal response rate (ORR)
Efficacy endpoint of CAR-BCMA T cells after infusion | through 24 months post administration of CAR-T-cells
  Complete Response (CR) /stringent Complete Response (sCR)
Efficacy endpoint of CAR-BCMA T cells after infusion | through 24 months post administration of CAR-T-cells
  ≥Very Good Partial Response (VGPR), including VGPR, CR, sCR
Efficacy endpoint of CAR-BCMA T cells after infusion | through 24 months post administration of CAR-T-cells
  Duration of Response (DOR)
Efficacy endpoint of CAR-BCMA T cells after infusion | through 24 months post administration of CAR-T-cells
  Clinical Benefit Rate (CBR)
Efficacy endpoint of CAR-BCMA T cells after infusion | through 24 months post administration of CAR-T-cells
  Time to Response (TTR)
Efficacy endpoint of CAR-BCMA T cells after infusion | through 24 months post administration of CAR-T-cells
  Minimal residual disease (MRD) negativity
Efficacy endpoint of CAR-BCMA T cells after infusion | through 24 months post administration of CAR-T-cells
  Progression Free Survival (PFS)
Efficacy endpoint of CAR-BCMA T cells after infusion | through 24 months post administration of CAR-T-cells
  Overall Survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Wenming CHEN, MD, Principal Investigator — Beijing Chao Yang Hospital; Zhengzheng FU, MD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (23):
- China (23):
  - The first affiliated hospital of bengbu medical college, Bengbu, Anhui
  - Beijing Chaoyang hospital, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Centre, Guangzhou, Guangdong
  - The 2nd People's Hospital of Shenzhen, Shenzhen, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The First Affiliated Hospital Of Soochow University, Suzhou, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The first Affiliated Hospital, College of medicine, Zhejiang University, Hanzhou, Zhejiang
  - The first Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Beijing Boren Hospital, Beijing
  - Beijing Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Tongji Hospital of Tongji University, Shanghai
  - Xinhua Hospital Affiliated To Shanghai Jiaotong University School of Medicine, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
  - Henan Provincial People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fu C, Chen W, Cai Z, Yan L, Wang H, Shang J, Wu Y, Yan S, Gao W, Shi X, Han X, Tang F, Zheng G, Wen Y, Meng X, Yuan D, Wang H, Li Z. Long-term follow-up of zevor-cel in patients with relapsed/refractory multiple myeloma. Blood Adv. 2026 Jan 27;10(2):468-478. doi: 10.1182/bloodadvances.2025017365. PMID 41160798